CLINICAL TRIAL: NCT03499990
Title: Prospective Study to Investigate Adrenal Crisis in Patients With Chronic Adrenal Insufficiency (Six-year Follow-up)
Brief Title: Study to Investigate Adrenal Crisis (Six-year Follow-up)
Status: Completed | Type: Observational
Sponsor: Wuerzburg University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: Adrenalcrisis-6FU
Record Dates: First submitted 2018-04-09; First posted 2018-04-17 (Actual); Last update posted 2018-04-18 (Actual); Status verified 2018-04

CONDITIONS: Adrenal Insufficiency
Keywords: Adrenal crisis; Risk factors
MeSH Terms: conditions — Adrenal Insufficiency

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Patients with adrenal insufficiency are at risk to suffer from life threatening adrenal crisis. The aim of this trial was to reevaluate the frequency of adrenal crisis and risk factors for crisis within a prospective study (six-years follow-up of a former prospective study).

DETAILED DESCRIPTION:
Despite established hormone replacement therapy, patients with chronic adrenal insufficiency are at risk of suffering from life threatening adrenal crisis with a considerable mortality. A former prospective study revealed a frequency of about 8 adrenal crisis/ 100 patient years and a crisis associated mortality of 0.5 per 100 patient years for patients; furthermore, patients with a previous adrenal crisis were at higher risk of crisis. The aim of the current trial was to reevaluate the frequency of adrenal crisis and risk factors by contacting the patients of the initial prospective study (see above) within a six-years follow-up. Patients are contacted by questionnaire and additionally by phone (in case of an adrenal crisis or implausible statements).

ELIGIBILITY:
Inclusion Criteria:

* Chronic primary or secondary adrenal insufficiency; hormone replacement therapy with glucocorticoids (hydrocortisone, cortisone acetat, prednisone or prednisolone)
* Written informed consent

Exclusion Criteria:

* Adrenal insufficiency due to adrenocortical carcinoma
* Adrenal insufficiency due to long-term pharmacological glucocorticoid treatment
* Glucocorticoid doses above 7.5 mg prednisolone equivalent for other reasons than adrenal insufficiency
* Age younger than 18 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Male and female patients with primary or secondary adrenal insufficiency that already participated in a former prospective study investigating adrenal crisis (Hahner et. al 2015).
Sampling Method: Non-Probability Sample
Enrollment: 268 (Actual)
Dates: Start 2016-08-13 (Actual); Primary Completion 2017-05-23 (Actual); Study Completion 2017-05-23 (Actual)

PRIMARY OUTCOMES:
Frequency of adrenal crisis | six years
  Evaluation of the frequency of adrenal crisis / number of adrenal crisis per patient years (adrenal crisis/100 patient years). Documentation of the number of adrenal crisis (within a follow-up-period of 6 years) of all participating patients.

SECONDARY OUTCOMES:
Risk factors | six years
  Identification of risk factors / confirmation of risk factors observed in former trials (previous adrenal crisis, female sex, diabetes insipidus) for adrenal crisis. Calculation of odds ratios.

REFERENCES:
- [Background] Hahner S, Spinnler C, Fassnacht M, Burger-Stritt S, Lang K, Milovanovic D, Beuschlein F, Willenberg HS, Quinkler M, Allolio B. High incidence of adrenal crisis in educated patients with chronic adrenal insufficiency: a prospective study. J Clin Endocrinol Metab. 2015 Feb;100(2):407-16. doi: 10.1210/jc.2014-3191. Epub 2014 Nov 24. PMID 25419882
- [Background] Hahner S, Loeffler M, Bleicken B, Drechsler C, Milovanovic D, Fassnacht M, Ventz M, Quinkler M, Allolio B. Epidemiology of adrenal crisis in chronic adrenal insufficiency: the need for new prevention strategies. Eur J Endocrinol. 2010 Mar;162(3):597-602. doi: 10.1530/EJE-09-0884. Epub 2009 Dec 2. PMID 19955259
- [Background] Smans LC, Van der Valk ES, Hermus AR, Zelissen PM. Incidence of adrenal crisis in patients with adrenal insufficiency. Clin Endocrinol (Oxf). 2016 Jan;84(1):17-22. doi: 10.1111/cen.12865. Epub 2015 Aug 27. PMID 26208266
- [Background] White K, Arlt W. Adrenal crisis in treated Addison's disease: a predictable but under-managed event. Eur J Endocrinol. 2010 Jan;162(1):115-20. doi: 10.1530/EJE-09-0559. Epub 2009 Sep 23. PMID 19776201